CLINICAL TRIAL: NCT04895722
Title: A Phase 2, Multicenter, Multi Arm, Study to Evaluate MK-1308A (Co-formulated Quavonlimab (MK-1308)/Pembrolizumab) Versus Other Treatments in Participants With Microsatellite Instability-High (MSI-H) or Mismatch Repair Deficient (dMMR) Stage IV Colorectal Cancer: (MK-1308A-008)
Brief Title: Evaluation of Co-formulated Pembrolizumab/Quavonlimab (MK-1308A) Versus Other Treatments in Participants With Microsatellite Instability-High (MSI-H) or Mismatch Repair Deficient (dMMR) Stage IV Colorectal Cancer (CRC) (MK-1308A-008/KEYSTEP-008)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1308A-008; MK-1308A-008 (Other: MSD); 2022-502100-70-00 (Other: EU CT); KEYSTEP-008 (Other: MSD); U1111-1283-2434 (Registry Identifier: UTN); 2020-005114-18 (EudraCT Number)
Record Dates: First submitted 2021-05-18; First posted 2021-05-20 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Colorectal Cancer
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Death-Ligand 1 (PDL1, PD-L1)
MeSH Terms: conditions — Colorectal Neoplasms; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Pembrolizumab (Active Comparator): Participants receive pembrolizumab 400 mg intravenously (IV) every 6 weeks (Q6W) for up to approximately 2 years.
  Interventions: Biological: Pembrolizumab
- Pembrolizumab/Quavonlimab (Experimental): Participants receive co-formulated pembrolizumab/quavonlimab (400 mg/25 mg) Q6W for up to approximately 2 years.
  Interventions: Biological: Pembrolizumab/Quavonlimab
- Pembrolizumab/Favezelimab (Experimental): Participants receive co-formulated pembrolizumab/favezelimab (200 mg/800 mg) every 3 weeks (Q3W) for up to approximately 2 years.
  Interventions: Biological: Pembrolizumab/Favezelimab
- Pembrolizumab/Vibostolimab (Experimental): Participants receive co-formulated pembrolizumab/vibostolimab (200 mg/200 mg) Q3W for up to approximately 2 years.
  Interventions: Biological: Pembrolizumab/Vibostolimab
- Pembrolizumab Plus MK-4830 (Experimental): Participants receive pembrolizumab 200 mg plus MK-4830 800 mg Q3W for up to approximately 2 years.
  Interventions: Biological: Pembrolizumab; Biological: MK-4830

INTERVENTIONS:
Biological: Pembrolizumab — 400 mg or 200 mg pembrolizumab administered via IV infusion.
  Other Names: MK-3475; Keytruda®
  Arms: Pembrolizumab; Pembrolizumab Plus MK-4830
Biological: Pembrolizumab/Quavonlimab — Co-formulated pembrolizumab/quavonlimab (400 mg/25 mg) fixed-dose combination (FDC) administered via IV infusion.
  Other Names: MK-1308A
  Arms: Pembrolizumab/Quavonlimab
Biological: Pembrolizumab/Favezelimab — Co-formulated pembrolizumab/favezelimab (200 mg/800 mg) FDC administered via IV infusion
  Other Names: MK-4280A
  Arms: Pembrolizumab/Favezelimab
Biological: Pembrolizumab/Vibostolimab — Co-formulated pembrolizumab/vibostolimab (200 mg/200 mg) FDC administered via IV infusion
  Other Names: MK-7684A
  Arms: Pembrolizumab/Vibostolimab
Biological: MK-4830 — 800 mg MK-4830 administered via IV infusion
  Arms: Pembrolizumab Plus MK-4830

SUMMARY:
The purpose of this study is to assess the efficacy and safety of co-formulated pembrolizumab/quavonlimab versus other treatments in participants with MSI-H or dMMR Metastatic Stage IV Colorectal Cancer.

ELIGIBILITY:
Inclusion Criteria:

* Has a histologically confirmed diagnosis of Stage IV CRC adenocarcinoma (as defined by American Joint Committee on Cancer [AJCC] version 8)
* Has locally confirmed dMMR/MSI-H
* Has a life expectancy of at least 3 months
* Female participants are eligible to participate if not pregnant or breastfeeding, and not a woman of childbearing potential (WOCBP), or if a WOCBP then uses a contraceptive method that is highly effective or is abstinent on a long-term and persistent basis, during the intervention period and for at least 120 days after the last dose of study intervention
* Has measurable disease per RECIST 1.1 as assessed by the site and verified by BICR
* Submit an archival (within 5 years of Screening) or newly obtained tumor tissue sample that has not been previously irradiated; formalin-fixed, paraffin embedded (FFPE) blocks are preferred to slides.
* Has adequate organ function

Cohort A:

- Has been previously treated for their Stage IV dMMR/MSI-H CRC and radiographically progressed on or after or could not tolerate standard treatment, which must include all of the following agents if approved and locally available in the country where the participant is randomized:

* Fluoropyrimidine, irinotecan and oxaliplatin (capecitabine is acceptable as equivalent to fluorouracil in prior therapy)
* With or without an anti-vascular endothelial growth factor (VEGF) monoclonal antibody (e.g., bevacizumab)
* At least one of the anti-epidermal growth factor receptor (EGFR) monoclonal antibodies (cetuximab or panitumumab) for rat sarcoma viral oncogene homolog (RAS) wild-type participants with left-sided tumors. Prior EGFR therapy is optional for patients with right sided RAS Wild-type (WT) tumors.

Cohort B:

- Has untreated Stage IV dMMR/MSI-H CRC with no prior chemotherapy or immunotherapy for this disease

Exclusion Criteria:

* Has received prior therapy with an agent directed to another stimulatory or coinhibitory T-cell receptor
* Has received prior systemic anticancer therapy including investigational agents within 4 weeks before the first dose of study intervention
* Has not recovered adequately from a surgery procedure, and/or has any complications from a prior surgery before starting study intervention
* Has received prior radiotherapy within 2 weeks of start of study intervention
* Has received a live or live-attenuated vaccine within 30 days before the first dose of study intervention
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks before the first dose of study intervention
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study medication
* Has a known additional malignancy that is progressing or has required active treatment within the past 2 years
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis
* Has severe hypersensitivity (≥Grade 3) to pembrolizumab, quavonlimab, favezelimab, vibostolimab, MK-4830, and/or any of their excipients
* Has an active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs)
* Has a history of (noninfectious) pneumonitis that required steroids or has current pneumonitis
* Has a history of acute or chronic pancreatitis
* Has neuromuscular disorders associated with an elevated creatine kinase
* Has urine protein ≥1 gram/24 hours
* Has an active infection requiring systemic therapy (e.g., tuberculosis, known viral or bacterial infections, etc.)
* Has a known history of Human Immunodeficiency Virus (HIV) infection
* Concurrent active Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] positive and/or detectable Hepatitis B Virus [HBV] deoxyribonucleic acid [DNA]) and Hepatitis C virus (defined as anti-HCV antibody positive and detectable HCV ribonucleic acid [RNA] infection
* Has clinically significant cardiac disease, including unstable angina, acute myocardial infarction within 6 months from Day 1 of study intervention administration, or New York Heart Association Class III or IV congestive heart failure. Medically controlled arrhythmia stable on medication is permitted.
* Has present or progressive accumulation of pleural, ascitic, or pericardial fluid requiring drainage or diuretic drugs within 2 weeks before randomization/allocation
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the treating investigator
* Has a known psychiatric or substance abuse disorder that would interfere with the participant's ability to cooperate with the requirements of the study
* Has had an allogenic tissue/solid organ transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2021-06-25 (Actual); Primary Completion 2025-05-21 (Actual); Study Completion 2026-06-25 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) as assessed by Blinded Independent Central Review (BICR) | Up to approximately 50 months
  ORR is defined as the percentage of participants who have a Complete Response (CR: disappearance of all target lesions) or a Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1. ORR as assessed by BICR will be presented.

SECONDARY OUTCOMES:
Duration of Response (DOR) per RECIST 1.1 as assessed by BICR | Up to approximately 50 months
  DOR is defined as the time from the first documented evidence of a CR (disappearance of all target lesions) or a PR (at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1 until Progressive Disease (PD) or death due to any cause, whichever occurs first, in participants demonstrating a CR or PR. Per RECIST 1.1, PD is defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD. DOR as assessed by BICR will be presented.
Progression-Free Survival (PFS) per RECIST 1.1 as assessed by BICR | Up to approximately 50 months
  PFS is defined as the time from randomization (or first dose) to the first documented PD per RECIST 1.1 or death from any cause, whichever occurs first. Per RECIST 1.1, PD is defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD. PFS as assessed by BICR will be presented.
PFS per RECIST 1.1 as assessed by Investigator | Up to approximately 50 months
  PFS is defined as the time from randomization (or first dose) to the first documented PD per RECIST 1.1 or death from any cause, whichever occurs first. Per RECIST 1.1, PD is defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD. PFS as assessed by investigator will be presented.
ORR per RECIST 1.1 as assessed by Investigator | Up to approximately 50 months
  ORR is defined as the percentage of participants who have a CR (disappearance of all target lesions) or a PR (at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1. ORR as assessed by investigator will be presented.
DOR per RECIST 1.1 as assessed by Investigator | Up to approximately 50 months
  DOR is defined as the time from the first documented evidence of a CR (disappearance of all target lesions) or a PR (at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1 until PD or death due to any cause, whichever occurs first, in participants demonstrating a CR or PR. Per RECIST 1.1, PD is defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD. DOR as assessed by investigator will be presented.
Overall Survival (OS) | Up to approximately 50 months
  OS is defined as the time from randomization (or first dose) to death due to any cause. OS will be presented.
Number of Participants Who Experienced an Adverse Event (AE) | Up to approximately 50 months
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study intervention. The number of participants with an AE will be presented.
Number of Participants Discontinuing Study Treatment Due to an AE | Up to approximately 50 months
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study intervention. The number of participants that discontinue study treatment due to an AE will be presented.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (109):
- United States (11):
  - Mid Florida Cancer Center ( Site 1519), Orange City, Florida
  - University Cancer & Blood Center, LLC ( Site 1521), Athens, Georgia
  - University of Chicago Medical Center-Medicine - Section of Hematology/Oncology - Gastrointestinal P, Chicago, Illinois
  - Icahn School of Medicine at Mount Sinai ( Site 1528), New York, New York
  - Hematology Oncology Associates of Rockland ( Site 1525), Nyack, New York
  - UPMC Hillman Cancer Center ( Site 1516), Pittsburgh, Pennsylvania
  - The West Clinic, PLLC dba West Cancer Center ( Site 1576), Germantown, Tennessee
  - Vanderbilt University Medical Center-Vanderbilt-Ingram Cancer Center ( Site 1509), Nashville, Tennessee
  - UT Southwestern Medical Center ( Site 1551), Dallas, Texas
  - Baylor Scott & White Medical Center - Temple-Division of Hematology/Oncology ( Site 1549), Temple, Texas
  - Northwest Medical Specialties, PLLC ( Site 1546), Tacoma, Washington
- Belgium (5):
  - UZ Brussel ( Site 0105), Brussels, Bruxelles-Capitale, Region de
  - Cliniques universitaires Saint-Luc-Medical Oncology ( Site 0104), Brussels, Bruxelles-Capitale, Region de
  - Université Catholique de Louvain-Namur - Centre Hospitalier -Oncology ( Site 0102), Yvoir, Namur
  - UZ Leuven ( Site 0101), Leuven, Vlaams-Brabant
  - AZ Delta vzw ( Site 0106), Roeselare, West-Vlaanderen
- Canada (3):
  - The Moncton Hospital-Oncology ( Site 0307), Moncton, New Brunswick
  - Sunnybrook Research Institute - Odette Cancer Centre ( Site 0316), Toronto, Ontario
  - McGill University Health Centre-CIM - Oncology ( Site 0306), Montreal, Quebec
- Colombia (7):
  - Instituto de Cancerología ( Site 1610), Medellín, Antioquia
  - Fundación Colombiana de Cancerología Clínica Vida ( Site 1606), Medellín, Antioquia
  - Clinica de la Costa S.A.S. ( Site 1608), Barranquilla, Atlántico
  - Clinica Colsanitas S.A, Sede Clínica Universitaria Colombia ( Site 1611), Bogotá, Bogota D.C.
  - Sociedad De Oncologia Y Hematologia Del Cesar-Oncology ( Site 1601), Valledupar, Cesar Department
  - Oncomédica S.A.S ( Site 1602), Montería, Departamento de Córdoba
  - Mediservis del Tolima IPS S.A.S ( Site 1609), Ibagué, Tolima Department
- Costa Rica (2):
  - CIMCA-Hemato-Oncology ( Site 2101), San José, Provincia de San José
  - Hospital Metropolitano - Sede Lindora-Metropolitano Research Institute Sede Lindora ( Site 2102), Santa Ana, Provincia de San José
- Denmark (4):
  - Rigshospitalet ( Site 1904), Copenhagen, Capital Region
  - Regionshospitalet Gødstrup ( Site 1901), Herning, Central Jutland
  - Aalborg Universitetshospital, Syd ( Site 1903), Aalborg, North Denmark
  - Odense Universitetshospital ( Site 1902), Odense, Region Syddanmark
- Estonia (2):
  - North Estonia Medical Centre Foundation-Chemotherapy ( Site 2301), Tallinn, Harju
  - Tartu University Hospital ( Site 2302), Tartu, Tartu
- France (6):
  - Assistance Publique Hôpitaux de Marseille - Hôpital de la Ti-Service d'Hepato-Gastro-Enterologie et, Marseille, Bouches-du-Rhone
  - Centre Georges François Leclerc ( Site 0506), Dijon, Cote-d Or
  - CHU Rangueil-Digestive oncology department ( Site 0502), Toulouse, Haute-Garonne
  - Hopital Claude Huriez - CHU de Lille ( Site 0510), Lille, Nord
  - Centre Hospitalier Universitaire de Poitiers ( Site 0511), Poitiers, Vienne
  - Hôpital Saint Antoine-Oncologie médicale ( Site 0508), Paris
- Germany (7):
  - Muenchen Klinik Neuperlach, Klinik fuer Haematologie und Onkologie ( Site 0612), Munich, Bavaria
  - Universitätsklinikum Marburg ( Site 0610), Marburg, Hesse
  - Kliniken Essen-Mitte, Evangelische Huyssens-Stiftung ( Site 0611), Essen, North Rhine-Westphalia
  - Universitaetsklinikum Carl Gustav Carus Dresden-Medical Dept I - Medical Oncology ( Site 0601), Dresden, Saxony
  - Otto-von-Guericke-Universität Magdeburg-Klinik für Gastroenterologie, Hepatologie und Infektiologie, Magdeburg, Saxony-Anhalt
  - Charité Universitaetsmedizin Berlin - Campus Mitte ( Site 0604), Berlin
  - Asklepios Altona-Oncology ( Site 0602), Hamburg
- Greece (4):
  - Alexandra General Hospital of Athens-ONCOLOGY DEPT. ( Site 2704), Athens, Attica
  - Evgenidion Hospital ( Site 2702), Athens, Attica
  - University General Hospital of Heraklion-Internal Medicine-Oncology ( Site 2703), Heraklion, Irakleio
  - European Interbalkan Medical Center-Oncology Department ( Site 2701), Thessaloniki
- Guatemala (5):
  - CELAN,S.A ( Site 2202), Guatemala City
  - INTEGRA Cancer Institute-Oncology ( Site 2201), Guatemala City
  - MEDI-K CAYALA ( Site 2205), Guatemala City
  - Centro Regional de Sub Especialidades Médicas SA ( Site 2204), Quetzaltenango
  - Centro Medico Integral De Cancerología (CEMIC) ( Site 2203), Quetzaltenango
- Hungary (6):
  - Pécsi Tudományegyetem Klinikai Központ-Onkoterápiás Intézet ( Site 2009), Pécs, Baranya
  - Bacs-Kiskun Megyei Korhaz-Onkoradiologiai Kozpont ( Site 2005), Kecskemét, Bács-Kiskun county
  - Jász-Nagykun-Szolnok Megyei Hetényi Géza Kórház-Onkologiai Kozpont ( Site 2001), Szolnok, Jász-Nagykun-Szolnok
  - Somogy Megyei Kaposi Mór Oktató Kórház-Oncology center ( Site 2010), Kaposvár, Somogy County
  - Semmelweis Egyetem-Belgyógyászati és Hematológiai Klinika ( Site 2002), Budapest
  - Debreceni Egyetem Klinikai Kozpont-Onkológiai Klinika ( Site 2008), Debrecen
- Italy (3):
  - Fondazione IRCCS Istituto Nazionale dei Tumori-Struttura Complessa Oncologia Medica 1 ( Site 0802), Milan, Lombardy
  - Istituto Nazionale Tumori IRCCS Fondazione Pascale-Department of Abdominal Oncology ( Site 0803), Napoli
  - Istituto Oncologico Veneto IRCCS ( Site 0804), Padua
- Lithuania (3):
  - Hospital of Lithuanian University of Health Sciences Kauno klinikos ( Site 2402), Kaunas, Kaunas County
  - National Cancer Institute ( Site 2401), Vilnius, Vilniaus Miestas
  - VILNIUS UNIVERSITY HOSPITAL SANTAROS KLINIKOS ( Site 2403), Vilnius
- Nederlands Kanker Instituut - Antoni van Leeuwenhoek (NKI-AVL) ( Site 2901), Amsterdam, North Holland, Netherlands
- Poland (6):
  - DOLNOSLASKIE CENTRUM ONKOLOGII PULMONOLOGII I HEMATOLOGII ( Site 0920), Wroclaw, Lower Silesian Voivodeship
  - Luxmed Onkologia sp. z o. o. ( Site 0915), Warsaw, Masovian Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - P-Klinika Onkologii i Radioterapii ( Site, Warsaw, Masovian Voivodeship
  - Mrukmed-Mrukmed ( Site 0901), Rzeszów, Podkarpackie Voivodeship
  - Szpital Wojewódzki im. Mikoaja Kopernika w Koszalinie-Oddzial Dzienny Chemioterapii ( Site 0903), Koszalin, West Pomeranian Voivodeship
  - Powiatowe Centrum Zdrowia ( Site 0911), Brzeziny, Łódź Voivodeship
- Romania (4):
  - Spitalul de Oncologie Monza Oncologie Medicala ( Site 2601), Bucharest, București
  - Fundeni Clinical Institute-Medical Oncology ( Site 2603), Bucharest, București
  - Cardiomed SRL Cluj-Napoca ( Site 2602), Cluj-Napoca, Cluj
  - Centrul de Oncologie "Sfântul Nectarie"-Medical Oncology ( Site 2604), Craiova, Dolj
- Russia (6):
  - Saint-Petersburg City Clinical Oncology Dispensary-Department of chemotherapy ( Site 1001), Saint Petersburg, Leningradskaya Oblast'
  - Fed State Budgetary Inst N.N. Blokhin Med Center of Oncology-Clinical Pharmacology and Chemotherapy, Moscow, Moscow
  - First Moscow State Medical University I.M. Sechenov-Interhospital Institution Health Management Cl, Moscow, Moscow
  - Rostov Cancer Research Institute ( Site 1014), Rostov-on-Don, Rostov Oblast
  - GBUZ SPb CRPCstmc(o) ( Site 1005), Saint Petersburg, Sankt-Peterburg
  - Republican Clinical Oncology Dispensary-Chemotherapy #3 ( Site 1006), Kazan', Tatarstan, Respublika
- South Korea (7):
  - Kyungpook National University Chilgok Hospital-Hematology/oncology ( Site 1103), Daegu, Taegu-Kwangyokshi
  - Korea University Anam Hospital ( Site 1107), Seoul
  - Seoul National University Hospital-Internal Medicine ( Site 1101), Seoul
  - Severance Hospital, Yonsei University Health System-Medical oncology ( Site 1104), Seoul
  - Asan Medical Center-Department of Oncology ( Site 1105), Seoul
  - Samsung Medical Center-Division of Hematology/Oncology ( Site 1102), Seoul
  - The Catholic Univ. of Korea Seoul St. Mary's Hospital-Medical Oncology ( Site 1106), Seoul
- Spain (8):
  - Hospital Universitario Marqués de Valdecilla ( Site 1202), Santander, Cantabria
  - Hospital Universitari Vall d'Hebron ( Site 1201), Barcelona, Catalonia
  - HOSPITAL GENERAL UNIVERSITARIO GREGORIO MARAÑON ( Site 1206), Madrid, Madrid, Comunidad de
  - H.R.U Malaga - Hospital General ( Site 1207), Málaga, Malaga
  - COMPLEJO HOSPITALARIO DE NAVARRA-oncologia médica ( Site 1210), Pamplona, Navarre
  - Hospital Universitario Central de Asturias-Medical Oncology ( Site 1203), Oviedo, Principality of Asturias
  - Fundación Instituto Valenciano de Oncología ( Site 1209), Valencia, Valenciana, Comunitat
  - Hospital Clinico San Carlos-Oncology Department ( Site 1204), Madrid
- Turkey (Türkiye) (5):
  - Baskent University Dr. Turgut Noyan Research and Training Center ( Site 1303), Adana
  - Hacettepe Universitesi-oncology hospital ( Site 1301), Ankara
  - Ankara City Hospital-Medical Oncology ( Site 1306), Ankara
  - Istanbul Universitesi Cerrahpasa-Medical Oncology ( Site 1302), Istanbul
  - TC Saglik Bakanligi Goztepe Prof. Dr. Suleyman Yalcin Sehir Hastanesi-oncology ( Site 1305), Istanbul
- United Kingdom (4):
  - Beatson West of Scotland Cancer Centre-Clinical Trials Unit ( Site 1401), Glasgow, Glasgow City
  - UCLH-Cancer Clinical Trials Unit ( Site 1402), London-Camden, London, City of
  - Velindre Cancer Centre-Research and Development ( Site 1415), Cardiff
  - University Hospital Coventry & Warwickshire ( Site 1406), Coventry

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- [Derived] Andre T, Pietrantonio F, Avallone A, Gumus M, Wyrwicz L, Kim JG, Yalcin S, Kwiatkowski M, Lonardi S, Zolnierek J, Odeleye-Ajakaye A, Leconte P, Fogelman D, Kim TW. KEYSTEP-008: phase II trial of pembrolizumab-based combination in MSI-H/dMMR metastatic colorectal cancer. Future Oncol. 2023 Dec;19(37):2445-2452. doi: 10.2217/fon-2022-1105. Epub 2023 Sep 13. PMID 37701986
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26204&tenant=MT_MSD_9011